CLINICAL TRIAL: NCT07293143
Title: Glycemic Effects of Meals - Repeatability Trial With Continuous Glucose Monitoring
Acronym: GEM-RT CGM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-46249
Record Dates: First submitted 2025-09-18; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Glucose Response
Keywords: Continuous glucose monitoring (CGM); Post prandial glucose; Fasting blood glucose; Hemoglobin (Hb)A1c; CGM-based dietary challenges; Metabolic risk

STUDY DESIGN:
Intervention Model Description: This is a pilot study where the order of the six study meals will be randomly assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Continuous glucose monitoring (Experimental): Each participant will have a Dexcom G6 CGM sensor applied to the upper arm. The order of the six study meals will be randomly assigned.
  Interventions: Other: Six meal challenges

INTERVENTIONS:
Other: Six meal challenges — Two of the meal challenges will only be provided once: (1) a 20oz bottle of Mountain Dew (2) a "typical breakfast" that participants would eat normally. The other four challenges consist of two meal events that will each be repeated: (1) two 8-ounce bottles of Ensure® nutritional shake (2) one cup of microwaved white rice (microwaveable Minute brand Jasmine Rice cups). The rice challenge will be performed once with normal chewing and once by swallowing without chewing, while the Ensure challenge will be repeated the same way on both days.

SUMMARY:
Almost half of adults in the United States have either diabetes mellitus (DM) or prediabetes (preDM), but many are undiagnosed and unaware of their condition. Current DM diagnosis and risk prediction are based on single "snapshot" measurements including: fasting blood glucose, postprandial glucose, and hemoglobin (Hb)A1c. Continuous glucose monitoring (CGM) offers a dynamic view of glucose levels throughout the day which enables characterizing individuals' dynamic glycemic profiles in response to physiological and environmental stimuli better than the conventional point-in-time glucose quantification approaches. By analyzing glycemic patterns from CGM tracings, it may be possible to identify individuals at increased risk of developing diabetes. However, an important prerequisite is to establish the reliability and consistency of glucose response patterns captured by CGM under controlled conditions.

Participants will be given six different meals to examine the glucose responses to these meals. Two of these meals (white rice and an Ensure drink) will be given twice for each participant to investigate whether individuals have the same glucose response to the same meal given on different days. Glucose will be measured using continuous glucose monitors, that have a thin wire sensor that measures glucose under the skin every five minutes for up to 10 days.

DETAILED DESCRIPTION:
This is a pilot study in which each participant undergoes six meal challenges (one each morning) under free-living conditions, while wearing a blinded CGM sensor. Glucose levels will be continuously measured, and meal challenge sequence will be randomly assigned to each participant.

The study objectives are to:

1. determine the within meal replicability of postprandial glucose response to a Ensure and White Rice meal challenges
2. evaluate if a whole food meal challenge (White Rice) exhibits lower reliability and greater physiological variability (under the chewing vs. not chewing condition) in postprandial glucose response compared to a standardized liquid mixed meal tolerance test (Ensure)
3. compare the postprandial average peak glucose response and 4 hour incremental area under the curve (iAUC) for the Ensure tolerance test, mountain dew tolerance test, White Rice, and typical breakfast.

These findings will inform the design of future studies and the potential use of CGM-based dietary challenges for early detection of metabolic risk.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy
* English speaking

Exclusion Criteria:

* Prior diagnosis of diabetes or taking medications that influence glucose metabolism, such as insulin, glucocorticoids, or Glucagon-like peptide-1 (GLP-1) receptor agonists.
* Taking hydroxyurea medication
* Taking beyond the maximum dose of acetaminophen (4g/day)
* Known food allergies or severe sensitivities to any study materials (dairy or soy)
* Limited and non-readers
* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Glycemic patterns from CGM | baseline, every 4 hours for 6 days
  Beginning at baseline, a 4-hour incremental area under the glucose curve (iAUC) will be calculated using the trapezoidal method. Peak glucose will be defined as the maximum glucose excursion within the 4-hour window. Continuous glucose monitoring (CGM) CGM values are recorded every 5 minutes, so linear interpolation will be used to provide a CGM value every minute to line up with the ingestion time documented in the participant's log.

SECONDARY OUTCOMES:
Fasting blood glucose levels | baseline, daily for 6 days
  This outcome will be assessed from the CGM data recorded after a10 hour fast.
Post prandial glucose levels | baseline, daily for 6 days
  This outcome will be assessed from the CGM data recorded daily 4 hours after a study meal.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole L Spartano, PhD, Principal Investigator — BUCA School of Medicine, Endocrinology, Diabetes, Nutrition and Weight Management

IPD SHARING:
Plan to Share IPD: No